CLINICAL TRIAL: NCT00178828
Title: Dynamic Measures of Neurochemistry in Mood Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000373; 5K23MH001828-03 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Depression; antidepressant; SSRI
MeSH Terms: conditions — Depression | interventions — Sertraline; Bupropion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: sertraline — Patients will be assigned by random selection to sertraline (50mg daily for one week, then 100mg daily) or bupropion (SR formulation, 150 mg daily for 1 week, then 150 mg BID). A second CSF collection will be completed after 4 weeks of the sertraline treatment (during week 5).
Drug: bupropion — Patients will be assigned by random selection to sertraline (50mg daily for one week, then 100mg daily) or bupropion (SR formulation, 150 mg daily for 1 week, then 150 mg BID). A second CSF collection will be completed after 4 weeks of the sertraline treatment (during week 5).

SUMMARY:
The purpose of this study is to understand changes in brain chemical signals when people take antidepressants called sertraline (Zoloft®) and bupropion (Wellbutrin SR, Zyban ®). Spinal fluid is used to measure chemical levels of dopamine, serotonin, and other chemicals thought to be involved in depression. The study has potential to help understand and treat depression.

DETAILED DESCRIPTION:
The purpose of this study is to understand changes in brain chemical signals when people take antidepressants called sertraline (Zoloft®) and bupropion (Wellbutrin SR, Zyban ®). Spinal fluid is used to measure chemical levels of dopamine, serotonin, and other chemicals thought to be involved in depression. The study has potential to help understand and treat depression.

ELIGIBILITY:
Inclusion Criteria:

* AGE RANGE: 18 to 50 years.
* WEIGHT: within 20% of ideal weight, as specified in the 1983 Metropolitan Height and Weight Tables. Patients who deviate from these ranges may be reviewed on an individual basis by the Investigator. This criterion is necessary because of mechanical risks of poor access in overweight individuals, and because of physiologic risks in underweight individuals.
* SEX DISTRIBUTION: both men and women (self or partner surgically sterilized, or using double barrier method). To the extent possible, women will have CSF sampling at the same point in their menstrual cycles, ideally during the follicular phase.
* RACE: any
* HEALTH: healthy, ambulatory depressed or healthy adults; must show clear capacity to form consent based on a strong understanding of the potential risks and benefits.

Exclusion Criteria:

* Evidence of significant hepatic, gastrointestinal, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular system abnormalities, history of deep venous thrombosis (DVT), thrombophlebitis, coagulopathy.
* Pregnancy.
* Patients with a known or suspected history of alcohol or drug misuse and/or a positive urine drug screen.
* Patients who are unwilling or unable to abide by the requirements of the study or who violate the prohibitions and restrictions of the study.
* Any condition which would make the patient, in the opinion of the Investigator, unsuitable for the study.
* Patients who have taken any unapproved prior or concomitant medications.
* Patients who have donated blood within one month of the study.
* Patients with serious medical illness, history or signs/symptoms of lumbar spine/disc disease or significant laboratory findings.
* Recent participation in other studies.
* Patients with histories of migraine will be considered individually, and warned of the risk of headache following spinal tap.
* Patients who smoke regularly, would experience withdrawal while hospitalized for 5 days, or who cannot abstain from tobacco for the entire duration of the study.
* Patients who present significant suicide risk, e.g. with a history of highly impulsive suicide attempts.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2002-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Power spectral density (PSD) of monoamine metabolite measures | Before antidepressant treatment and after 4 weeks of antidepressant treatment (during week 5)
  Power spectral density measures the rhythmicity, or periodicity, of the time series of monoamine metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Salomon, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States